CLINICAL TRIAL: NCT00129805
Title: Sarpogrelate-Aspirin Comparative Clinical Study for Efficacy and Safety in Secondary Prevention of Cerebral Infarction (S-ACCESS): A Randomized, Double-Blind, Aspirin-Controlled Trial
Brief Title: Sarpogrelate-Aspirin Comparative Clinical Study for Efficacy and Safety in Secondary Prevention of Cerebral Infarction (S-ACCESS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: General Manager, Clinical Research Department I, Mitsubishi Tanabe Pharma Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MCI9042-15
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2008-08

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — sarpogrelate; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCI-9042 (Experimental)
  Interventions: Drug: MCI-9042
- Aspirin (Active Comparator)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: MCI-9042
  Other Names: Sarpogrelate(INN); ANPLAG(R)
  Arms: MCI-9042
Drug: Aspirin
  Arms: Aspirin

SUMMARY:
Sarpogrelate (MCI-9042) is an antiplatelet drug that decreases 5-hydroxytryptamine (5-HT) levels in platelets via a blockade of 5-HT2 receptors; it has been used in atherosclerotic peripheral arterial disease.

S-ACCESS was a randomized, double-blinded trial to compare the relative efficacy of sarpogrelate (100mg three times daily) and aspirin (81mg once daily) in 1510 patients with recent cerebral infarction. Patients were followed for 0.9 to 3.5 years. The primary endpoint was recurrence of cerebral infarction; relative safety was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral infarction except cardiac source of embolism
* Onset ≧ 1 week to ≦ 6 months before randomization
* Neurological signs persisting ≧ 1 day from onset
* Computed tomography (CT) or magnetic resonance imaging (MRI) detection of responsible site
* Age ≧ 20 years
* Systolic pressure ≦ 180 mmHg; diastolic pressure ≦ 110 mmHg

Exclusion Criteria:

* Functional outcome at randomization: Modified Rankin Scale = 4, 5
* Previous or planned vascular surgery for cerebral infarction
* History of intracranial hemorrhage
* History of systemic bleeding, or other history of bleeding diathesis or coagulopathy
* Severe complications (renal or hepatic insufficiency, heart failure, hemopathy, etc.)
* Pregnant or possibly pregnant women, or nursing mothers
* History of sarpogrelate and aspirin sensitivity
* Treating malignant tumor or treated within 5 years
* Current peptic ulceration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1510 (Actual)
Dates: Start 2001-01; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
recurrence of cerebral infarction

SECONDARY OUTCOMES:
intracerebral hemorrhage, subarachnoid hemorrhage, undetermined stroke, transient ischemic attack, myocardial infarction, unstable angina, or vascular death

CONTACTS AND LOCATIONS:
Overall Officials: Yukito Shinohara, MD, Study Chair — Federation of National Public Service Personnel Mutual Aid Associations Tachikawa Hospital

REFERENCES:
- [Result] Shinohara Y, Nishimaru K, Sawada T, Terashi A, Handa S, Hirai S, Hayashi K, Tohgi H, Fukuuchi Y, Uchiyama S, Yamaguchi T, Kobayashi S, Kondo K, Otomo E, Gotoh F; S-ACCESS Study Group. Sarpogrelate-Aspirin Comparative Clinical Study for Efficacy and Safety in Secondary Prevention of Cerebral Infarction (S-ACCESS): A randomized, double-blind, aspirin-controlled trial. Stroke. 2008 Jun;39(6):1827-33. doi: 10.1161/STROKEAHA.107.505131. Epub 2008 Apr 3. PMID 18388340